CLINICAL TRIAL: NCT03673163
Title: Lidocaine Infusion for Pain After Herniotomy (LIPAH), A Randomized Placebo-controlled Trial (LIPAH Trial)
Brief Title: Lidocaine Infusion for Pain After Herniotomy
Acronym: LIPAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Xiangcai Ruan, MD, PhD, Vice-Director in Dept Anesth & Pain, Professor, Guangzhou First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GZFPH-2018-115
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Hernia, Inguinal; Lidocaine; Pain, Postoperative; Chronic Pain
Keywords: chronic postoperative pain; lidocaine infusion; inguinal herniotomy
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Chronic Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental): Lidocaine treatment
  Interventions: Drug: Lidocaine
- Control (Placebo Comparator): Placebo treatment
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Lidocaine — Infusion of 2% lidocaine hydrochloride at 4 mL/h,prior to surgery and discontinued until 24 h after surgery.
  Other Names: intravenous lidocaine infusion
  Arms: Lidocaine
Drug: Control — Infusion of normal saline at 4 mL/h, prior to surgery and discontinued until 24 h after surgery.
  Other Names: normal saline control
  Arms: Control

SUMMARY:
This study seeks to investigate lidocaine infusion to reduce occurrence of chronic postoperative pain at 3-month after inguinal herniotomy

DETAILED DESCRIPTION:
Inguinal hernia repair is associated with a 5%-30% incidence of chronic pain; however, the pathogenesis remains unknown, and few studies have assessed chronic pain as the primary aim of the study. Lidocaine infusion could be a possible approach to reducing the prevalence of chronic pain after herniotomy. Recently, a meta-analysis concluded a modest but statistically significant reduction of pain severity in the first four postoperative hours measured by the visual analogue scale (mean difference, -0.84; 95% CI, -1.10 to -0.59). However, a more recent meta-analysis found that only limited clinical data and biological plausibility support lidocaine infusions for the prevention of postoperative persistent pain (odds ratio, 0.29; 95% CI, 0.18 to 0.48). This study was designed to investigate whether lidocaine infusion after inguinal herniotomy would lower the incidence of chronic postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo unilateral inguino herniotomy

Exclusion Criteria:

* (1)ASA classification status III or above
* (2)Body weight<35kg
* (3)Liver cirrhosis
* (4)A history of previous herniotomy
* (5)Pregnancy
* (6)Severe arrhythmia
* (7)Congestive heart failure
* (8)Opioid or steroid use 6 months before surgery
* (9)Allergy to lidocaine
* (10)Chronic pain syndrome (any type)
* (11)Emergency surgery
* (12)Incapacity to give an informed consent, Visual dysfunction or severe mental disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of chronic pain | At 3 months after surgery.
  Chronic pain was assessed in accordance with the IMMPACT recommends in the domains of: (1) absence or presence of pain in the area of the surgery, (2) clinically important (NRS ≥ 4 on a 0- to 10-point scale) daily average pain, (3) clinically important pain at rest, (4) clinically important pain intensity upon movement or activity, (5) pain qualities, and (6) physical and emotional functioning.

SECONDARY OUTCOMES:
Postoperative acute pain | Up to 48 hours after surgery
  Use an 11-point Numeric Rating Scale (NRS) to assess the postoperative acute pain
Sedation | Up to 48 hours after surgery
  Use an 0- to 10-point Numeric Rating Scale to asses
Postoperative nausea and vomiting (PONV) | Up to 48 hours after surgery
  Use an 0- to 10-point Numeric Rating Scale to asses
Fatigue | Up to 48 hours after surgery
  Use an 0- to 10-point Numeric Rating Scale to asses
Chronic pain at 6-month after surgery | At 6 months after surgery.
  Chronic pain was assessed in accordance with the IMMPACT recommends in the domains of: (1) absence or presence of pain in the area of the surgery, (2) clinically important (NRS ≥ 4 on a 0- to 10-point scale) daily average pain, (3) clinically important pain at rest, (4) clinically important pain intensity upon movement or activity, (5) pain qualities, and (6) physical and emotional functioning.
Chronic pain at 12-month after surgery | At 12 months after surgery.
  Chronic pain was assessed in accordance with the IMMPACT recommends in the domains of: (1) absence or presence of pain in the area of the surgery, (2) clinically important (NRS ≥ 4 on a 0- to 10-point scale) daily average pain, (3) clinically important pain at rest, (4) clinically important pain intensity upon movement or activity, (5) pain qualities, and (6) physical and emotional functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcai Ruan, PhD, Principal Investigator — Affliated First People's Hospital of Guangzhou ,Guangzhou Medical University
Locations (1):
- Guangzhou First People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang JL, Zhang WJ, Gao M, Zhang S, Tian DH, Chen J. A cross-cultural adaptation and validation of the short-form McGill Pain Questionnaire-2: Chinese version in patients with chronic visceral pain. J Pain Res. 2017 Jan 5;10:121-128. doi: 10.2147/JPR.S116997. eCollection 2017. PMID 28115872
- [Background] Kranke P, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Weibel S. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery. Cochrane Database Syst Rev. 2015 Jul 16;(7):CD009642. doi: 10.1002/14651858.CD009642.pub2. PMID 26184397
- [Background] Bailey M, Corcoran T, Schug S, Toner A. Perioperative lidocaine infusions for the prevention of chronic postsurgical pain: a systematic review and meta-analysis of efficacy and safety. Pain. 2018 Sep;159(9):1696-1704. doi: 10.1097/j.pain.0000000000001273. PMID 29757886
- [Background] Dworkin RH, Turk DC, Peirce-Sandner S, Baron R, Bellamy N, Burke LB, Chappell A, Chartier K, Cleeland CS, Costello A, Cowan P, Dimitrova R, Ellenberg S, Farrar JT, French JA, Gilron I, Hertz S, Jadad AR, Jay GW, Kalliomaki J, Katz NP, Kerns RD, Manning DC, McDermott MP, McGrath PJ, Narayana A, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Reeve BB, Rhodes T, Sampaio C, Simpson DM, Stauffer JW, Stucki G, Tobias J, White RE, Witter J. Research design considerations for confirmatory chronic pain clinical trials: IMMPACT recommendations. Pain. 2010 May;149(2):177-193. doi: 10.1016/j.pain.2010.02.018. Epub 2010 Mar 6. PMID 20207481
- [Background] Aasvang E, Kehlet H. Chronic postoperative pain: the case of inguinal herniorrhaphy. Br J Anaesth. 2005 Jul;95(1):69-76. doi: 10.1093/bja/aei019. Epub 2004 Nov 5. No abstract available. PMID 15531621